CLINICAL TRIAL: NCT05383404
Title: Clinical and Laboratory Parameters Associated With Different Degrees of Dehydration Among Children With Diabetic Ketoacidosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Ismail, resident doctor at pediatric department at faculty of medicine sohag university hospital, Sohag University
Other Study IDs: Soh-Med-22-05-11
Record Dates: First submitted 2022-05-16; First posted 2022-05-20 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetic Ketoacidosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mild dehydration: (3-5)% according to change in body weight.
  Interventions: Diagnostic Test: blood and urine samples
- moderate dehydration: (6-9)% according to change in body weight.
  Interventions: Diagnostic Test: blood and urine samples
- severe dehydration: (6-9)% according to change in body weight.
  Interventions: Diagnostic Test: blood and urine samples

INTERVENTIONS:
Diagnostic Test: blood and urine samples — complete blood count, blood glucose, blood gases, serum bicarbonates, serum electrolytes, serum albumin ,serum creatinine. blood urea nitrogen, urine analysis.

SUMMARY:
Diabetic ketoacidosis (DKA) is a common acute complication of type 1 diabetes mellitus (T1DM). DKA is characterized by hyperglycemia, metabolic acidosis, increased levels of ketone bodies in blood and urine. This leads to osmotic diuresis and severe depletion of water and electrolytes from both the intra- and extracellular fluid (ECF) compartments.

Estimation of the degree of dehydration for children admitted with DKA is of great clinical importance. The calculation of the amount of deficit therapy depends on the estimated degree of dehydration. However, the degree of dehydration present during DKA is difficult to be clinically assessed. Hyperosmolality tends to preserve intravascular volume with maintenance of peripheral pulses, blood pressure, and urine output until extreme volume depletion occurs. Metabolic acidosis leads to hyperventilation and dry oral mucosa as well as decreased peripheral vascular resistance and cardiac function . consequently, hyper-osmolality may lead to an underestimation of the degree of dehydration, whereas metabolic acidosis may lead to an overestimation of the degree of dehydration. This makes the physical findings unreliable in this setting.

Several clinical and biochemical markers were suggested to assess and stage the degree of dehydration at hospital admission. The blood urea nitrogen , hematocrit , plasma albumin are useful markers of the degree of ECF contraction.However, Several previous studies demonstrated that there was no agreement between assessed and measured degree of dehydration which is calculated according to change in body weight at admission and after correction of dehydration. there were tendencies to overestimated or underestimate the degree of dehydration between different physicians. The assessment of the magnitude of dehydration in DKA is of major interest and continues to be a subject of research.

This study aims to assess the association between different clinical and laboratory parameters in children with diabetic ketoacidosis and the degree of dehydration at hospital admission among those children.

ELIGIBILITY:
Inclusion Criteria:

* Children with T1DM aged 0-12 years admitted to the pediatric emergency department with DKA criteria (blood glucose level > 200 mg/dl, pH < 7.3, and /or bicarbonate level in blood < 15 mmol/l and positive ketones in urine by dipstick method) will be included.

Exclusion Criteria:

* Children with DKA who are referred to Sohag university hospital after starting treatment for DKA at another hospital.

Ages: 1 Hour to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with T1DM aged 0-12 years admitted to the pediatric emergency department with DKA criteria (blood glucose level > 200 mg/dl, pH < 7.3, and /or bicarbonate level in blood < 15 mmol/l and positive ketones in urine by dipstick method) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-25 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
measured degree of dehydration | 1year
  calculated as percentage of the difference between the weight at disharge from Picu and the weight at admission to the weight at disharge from Picu

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vicinanza A, Messaaoui A, Tenoutasse S, Dorchy H. Diabetic ketoacidosis in children newly diagnosed with type 1 diabetes mellitus: Role of demographic, clinical, and biochemical features along with genetic and immunological markers as risk factors. A 20-year experience in a tertiary Belgian center. Pediatr Diabetes. 2019 Aug;20(5):584-593. doi: 10.1111/pedi.12864. Epub 2019 May 15. PMID 31038262
- [Background] Raghupathy P. Diabetic ketoacidosis in children and adolescents. Indian J Endocrinol Metab. 2015 Apr;19(Suppl 1):S55-7. doi: 10.4103/2230-8210.155403. PMID 25941653
- [Background] Ugale J, Mata A, Meert KL, Sarnaik AP. Measured degree of dehydration in children and adolescents with type 1 diabetic ketoacidosis. Pediatr Crit Care Med. 2012 Mar;13(2):e103-7. doi: 10.1097/PCC.0b013e3182231493. PMID 21666534
- [Background] Wolfsdorf JI, Glaser N, Agus M, Fritsch M, Hanas R, Rewers A, Sperling MA, Codner E. ISPAD Clinical Practice Consensus Guidelines 2018: Diabetic ketoacidosis and the hyperglycemic hyperosmolar state. Pediatr Diabetes. 2018 Oct;19 Suppl 27:155-177. doi: 10.1111/pedi.12701. No abstract available. PMID 29900641